CLINICAL TRIAL: NCT05273255
Title: An Open Label Feasibility Study of Fecal Microbiota Transplantation (FMT) in Patients With Malignancies Not Responding to Cancer Immunotherapy (CI)
Brief Title: Fecal Microbiota Transplantation in Patients With Malignancies Not Responding to Cancer Immunotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Scharl (Other)
Responsible Party: Sponsor-Investigator, Michael Scharl, Prof. Dr. med., University of Zurich
Organization: University of Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FMT-Malignancies
Record Dates: First submitted 2022-02-14; First posted 2022-03-10 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Fecal Microbiota Transplantation; Immune Checkpoint Inhibitors; Immunotherapy
MeSH Terms: conditions — Neoplasms | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMT-Recipients (Experimental): FMT-Recipients are patients with stage IV cancer, who have not sufficiently responded (stable disease or non-response) after at least 1 full cycle of CI. These patients will undergo the FMT procedure after the colon cleansing performed per routine treatment protocols at the Departement of Gastroenterology at the University Hospital of Zürich.
  The stool is donated by FMT-Donors, which are patients with any solid cancer stage III or IV cancers, who received any ICI-Therapy and have experienced a durable partial or complete response.
  FMT infusate will be administered via colonoscopy.
  Interventions: Biological: Fecal Microbiota Transplantation (FMT)

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation (FMT) — Single-dose of fecal microbiota from FMT-Donor transplanted endoscopically to FMT-Recipient in between two cycles of CI.

SUMMARY:
The intestinal microbiome forms a symbiotic relationship with the human host and continuously interacts with its immune system. Specific compositions of the intestinal microbiome in patients with cancer have been linked to the response to therapy with cancer immunotherapies (CI), such as immune checkpoint inhibitors (ICIs). The investigators hypothesize that fecal microbiota transplantation (FMT) from patients being responsive to ICI therapy (FMT-Donor) can modulate the intestinal microbiome of patients with CI-refractory malignancies (FMT-Recipients) and render them into responders. Successful proof-of-concept studies showed that reversion from an ICI non-responsive to a responsive disease is indeed possible in melanoma patients after FMT. This trial expands the FMT intervention to patients with any malignancy treated with cancer immunotherapy as a standard of care, to demonstrate the feasibility of this FMT approach as a novel option in cancer therapy.

ELIGIBILITY:
General inclusion criteria for all participants:

* Patients, at minimum 18 years of age, male or female
* Signed informed consent obtained from subject according to local regulations
* ECOG score at the time of study enrolment 0-1

The investigators will include patients/individuals fulfilling inclusion criteria for one of the following groups:

1. Patients with refractory malignancy (FMT-Recipients). The investigators will recruit 25 individuals with stable or progressing disease after minimum of 1 cycle of CI.
2. Patients with malignancy in remission after ICI therapy (FMT-Donors). The investigators will recruit 5 patients willing to donate stool samples for the study.

Inclusion criteria FMT-Recipients:

1. Histologically or cytologically confirmed diagnosis of malignancy
2. Currently treated with CI with at least 1 cycle completed. Multiple active malignancies are allowed.
3. Patient with stable or progressive disease as shown at the most recent staging method and decided by the treating investigator (based on the radiologic assessment).
4. Must be CI refractory/resistant as judged by the treating physician based on a recent CT or PET-CT (PET-MRI) scan not older than 8 weeks before screening visit.
5. Willingness to receive FMT administered via colonoscopy and undergo necessary bowel preparation pre-procedure.
6. Demonstrate adequate organ function as defined below, all screening labs should be performed within 28 days of FMT intervention.

   Following laboratory parameters need to be met:
   * Platelet count ≥ 50 x 10^9 / L
   * Hemoglobin ≥ 8.5 g/dL
   * Prothrombin time (PT)-international normalized ration (INR) ≤ 1.5
7. Female subject of childbearing potential should have a negative urine pregnancy within minimum 8 hours prior to receiving the study intervention (FMT). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
8. Female subjects of childbearing potential must be willing to use a clinically established method of contraception before the FMT procedure.

Inclusion criteria FMT-Donors:

1. Documented history of malignancy treated with ICI therapy.
2. Featuring partial or complete response of the malignancy as assessed by radiologic examination with a minimum duration of remission lasting ≥12 months measured since initiation of therapy.
3. Willingness to complete donor-specific questionnaire.
4. Willingness to complete donor-specific serologic and stool testing to evaluate infectious agents.
5. Patient tested negatively for all infectious agents specified.
6. Willingness to provide multiple stool samples, until total amount reaches 170g.
7. Absence of major gastrointestinal symptoms 3 months prior to stool donation (including frequent vomiting, diarrhea, bleeding, constipation).

Exclusion criteria FMT Recipients:

1. Presence of absolute contra-indications to colonoscopy and/or FMT administration:

   * Toxic megacolon
   * Inflammatory bowel disease
   * Anatomic contra-indications to colonoscopy
   * Colectomy
2. Patient is currently participating and receiving other study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of this study intervention.
3. Currently under any form of systemic antibiotics.
4. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (> 10 mg prednisone daily or equivalent) or any other form of immunosuppressive therapy two weeks prior to trial treatment. Patients receiving systemic steroids at physiologic doses are permitted to enroll assuming steroid dose is not above the acceptable threshold (> 10 mg prednisone daily or equivalent).
5. Severe anaphylactic reaction to any food (food allergies).
6. Had a severe hypersensitivity reaction to propofol.
7. Has serious concomitant illnesses. The eligibility can be granted by the treating investigator on individual bases.
8. Has HIV infection or AIDS-related illness.
9. Has active infection of HAV, HBV or HCV. Patients with a history of Hepatitis B/C infection who have received anti-viral therapy and are disease free may be considered for enrollment after discussion with Principal Investigator.
10. Patient has received a live vaccine within 4 weeks prior to the first dose of treatment. Seasonal influenza vaccines or COVID-19 vaccines for injection are generally inactivated virus vaccines and are allowed.
11. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
12. Females who are pregnant or breastfeeding.
13. Active central nervous system (CNS) metastases and/or leptomeningeal involvement.

Exclusion criteria FMT Donors:

1. History or current antibiotic treatment during the 2 month preceding donation.
2. History or current intrinsic gastrointestinal illnesses, including inflammatory bowel disease, irritable bowel syndrome, chronic diarrheal disorder (e.g. celiac disease or microscopic colitis) or major gastrointestinal surgical procedures.
3. History or current symptomatic autoimmune illness.
4. History or current documented neurologic or neurodevelopmental disorders.
5. History or current metabolic syndrome, obesity (BMI of >35), or moderate-to-severe malnutrition (as assessed clinically).
6. History or current infection with HIV (or AIDS-related illness).
7. Positive serological tests for Syphilis, HAV, HBV or HCV.
8. Positive stool test for Escherichia coli, Vancomycin-resistant Enterococcus, Norovirus, C. difficile, Yersinia, Campylobacter, Shigella or Salmonella.
9. Positive stool test for parasites.
10. Positive Sars-CoV-2 screening/testing (active infection).

Subjects whose pregnancy test on Screening visit shows a positive result, have to be excluded from the study. All pregnancies occurring during the treatment phase of the study and within 30 days after discontinuation of study medication have to be reported to the Investigator-Sponsor within one working day of the investigational sites knowledge of the pregnancy on the Initial Pregnancy Report Form. Female Subjects should be informed in this way before signing the informed consent form. Female partners of male participants may get pregnant without any consequence to the male participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Change in the intestinal microbiome community | up to 24 weeks
  Mean change from baseline of bacterial species compared with 24 weeks post fecal microbiota transplantation (FMT).

SECONDARY OUTCOMES:
Adverse Events Related to Study Intervention | up to 24 weeks
  Number of adverse events and serious adverse events related definitely to fecal microbiota transplantation (FMT).
Objective Response Rate | up to 24 weeks
  Percentage of participants that achieved an objective response as per Response Evaluation Criteria in Solid Tumours (iRECIST) treated with immunotherapy.
Progression-Free Survival | up to 24 weeks
  Time, measured in days, between the fecal microbiota transplantation (FMT) and disease progression as per Response Evaluation Criteria in Solid Tumours (iRECIST) treated with immunotherapy.
Overall Survival | up to 24 weeks
  The length of time (in days) from study intervention that participants remain alive.
Correlation between specific immune cell presence in blood/colon tissue and therapy response | up to 24 weeks
  Number of immune cells in peripheral blood, intestinal and tumor tissue at the time of stool donation, baseline and after 24 weeks post fecal microbiota transplantation (FMT).
CI response rate upon microbiome change | up to 24 weeks
  Number of participants with specific bacteria species that positively correlate with the favorable response to cancer immunotherapy.
Quality of life based on the questionnaire | up to 24 weeks
  Scoring based on "European Organization for Research and Treatment of Cancer 30-item quality of life questionnaire (EORTC QLQ C-30)".

CONTACTS AND LOCATIONS:
Overall Officials: Michael Scharl, Prof. Dr., Principal Investigator — University Hospital Zurich, University of Zurich
Locations (1):
- University of Zurich, University Hospital Zurich, Zurich, Switzerland